CLINICAL TRIAL: NCT05549596
Title: A Single-center, Open-label, Randomized, Parallel-group, Standard Therapy Controlled, Equivalence Clinical Trials to Evaluate the Efficacy and Safety of Structural Changes in the Spine to Determine the Traction Effect of an Investigational Device, Ceragem Master V6 (CGM MB-1701) Use in Patients With Lumber Disc Herniation & Degenerative Spinal Stenosis
Brief Title: CETIS-I (CEra Traction Improves Spine-I)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceragem Clinical Inc. (Industry)
Responsible Party: Sponsor
Organization: Ceragem Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC_MV6_208
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lumbar Disc Herniation; Degenerative Spinal Stenosis; Spine Traction
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traction treatment (Experimental): About 40 minutes spine traction including temperature application, Spine Scan, Pre-stroke, and Main Stroke
  Interventions: Device: Ceragem Master V6 Traction
- Physical Therapy (Active Comparator): About 40 minutes standard physical therapy including temperature application and traction
  Interventions: Device: Physical therapy with standard traction device

INTERVENTIONS:
Device: Ceragem Master V6 Traction — Ceragem Master V6 Traction for L2~L3
  Arms: Traction treatment
Device: Physical therapy with standard traction device — Physical therapy with standard traction device
  Arms: Physical Therapy

SUMMARY:
In this clinical trial, equivalence is evaluated by exploratory comparison of changes in X-Ray lesions with test group (Cerazem Master V6) and control group (physical therapy) in patients with intervertebral disc herniation and degenerative stenosis.

DETAILED DESCRIPTION:
The efficacy and safety evaluation are conducted before and after the application of the test device. The investigator shall apply an investigational device once when visiting a suitable subject for one day (Arm;Traction treatment) or standard physical therapy including temperature application and traction(Arm;Physical Therapy)

ELIGIBILITY:
Inclusion Criteria:

* Subject who has been diagnosed with intervertebral disc herniation or degenerative stenosis (a person who has been diagnosed in the past or has been diagnosed upon obtaining consent)
* Adult men and women over 19 years of age
* Body mass index (BMI) 18.5 over to less than 30

Exclusion Criteria:

* Subject with fibromyalgia, dystonia, and epilepsy
* Subject with sensory impairment
* Subject with physical irritation-induced skin lesions such as fever and compression (dermatosis, compression urticaria, choline urticaria, fever urticaria, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Anterior and posterior distance changes of L2-S1 intervertebral disc | Immediately after application
  Anterior and posterior distance changes of L2-S1 intervertebral disc are evaluated through X-Ray immediately after application of medical device compared to baseline

SECONDARY OUTCOMES:
Ratio of L2-S1 Anterior/posterior intervertebral distance | Immediately after application
  Ratio of L2-S1 Anterior/posterior intervertebral distance evaluated by X-Ray immediately after application of medical device compared to baseline (A/P ratio)
Changes in lower extremity radiation pain | Immediately after application
  Changes in lower extremity radiation pain evaluated through VAS immediately after application of medical device compared to baseline
Changes in the range of waist movement | Immediately after application
  Changes in the range of waist movement evaluated by the Schober test immediately after one application of medical device compare to baseline
Change in the angle evaluated by the SLR test | Immediately after application
  Change in the angle evaluated by the Straight Leg Rasing test (SLR test) modified immediately after the application of the medical device compared to the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yong Soon Yoon, Principal Investigator — Presbyterian Medical Cente
Locations (1):
- Presbyterian Medical Center, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No